CLINICAL TRIAL: NCT06264401
Title: Treatment Exercises With Core Stability and Dynamic Resistance Exercise for Postmenopausal Women With Osteoporosis: A Randomized Controlled Trial
Brief Title: Treatment Exercises With Core Stability and Dynamic Resistance Exercise for Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen Shaaban Abd El Azeim, principle investgator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: menopausal with osteoporsis
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Postmenopausal Osteoporosis
Keywords: postmenopausal; osteoporosis; corestability; dynamic resistance; bone mineral density
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Intervention Model Description: intervention: medication the experimental and control groups received (Alendronate) 70 mg 1 tab every week for 4 months.
  treatment exercises the experimental group performed core stability and dynamic resistance exercises, a 45-min lumbar-pelvic/core strength and stability exercise program which include 5 min warming up and 5 min cooling down at the end of the session each exercise was executed for three sets of 15 seconds, which gradually upgraded to three sets of 45-second at the fourth month and 10 sec rest between each set and dynamic resistance exercise performed by each woman for 2 sets for 8-12 repetitions gradually along the study of 90 sec rest between each set for a duration of 60 min including 10 min warming up and 10 min cooling down in form of stretching.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placepo group (Experimental): Alendronate:
  the experimental and control group received (Alendronate) 70 mg 1 tab every week for 4 months.
  Interventions: Other: Alendronate
- exercises and alendronate group (Experimental): alendronate: the experimental and control group received (Alendronate) 70 mg 1 tab every week for 4 months.
  treatment exercises: the experimental group performed core stability and dynamic resistance exercises, a 45-min lumbar-pelvic/core strength and stability exercise program which include 5 min warming up and 5 min cooling down at the end of the session each exercise was executed for three sets of 15 seconds, which gradually upgraded to three sets of 45-second at the fourth month and 10 sec rest between each set and dynamic resistance exercise performed by each woman for 2 sets for 8-12 repetitions gradually along the study of 90 sec rest between each set for a duration of 60 min including 10 min warming up and 10 min cooling down in form of stretching.
  Interventions: Other: Alendronate; Other: treatment exercises

INTERVENTIONS:
Other: Alendronate — control group received (Alendronate) 70 mg 1 tab every week.
Other: treatment exercises — the experimental group performed core stability and dynamic resistance exercises, a 45-min lumbar-pelvic/core strength and stability exercise program, each exercise was executed for three sets of 15 seconds, which gradually upgraded to three sets of 45-second at the fourth month and 10 sec rest between each set and dynamic resistance exercise performed by each woman for 2 sets for 8-12 repetitions gradually along the study of 90 sec rest between each set for a duration of 60 minutes.
  Arms: exercises and alendronate group

SUMMARY:
osteoporosis is a common disease that affect most of postmenopausal women. various treatment procedures are used to avoid future complain among postmenopausal population.

DETAILED DESCRIPTION:
Ethics statement This study was approved by the institutional review board of the faculty of physical therapy, Cairo university, Egypt (no.P.T. REC/012/003867) and strictly adhered to the criteria proclaimed in the latest version of the declaration of Helsinki code of ethics. each woman freely consents to participate in this research study.

study design. A prospective double-masked randomized controlled trial.

sample size calculation. Based on a pilot study, sample size was calculated according to the significant difference in the value of mean difference (pretreatments - posttreatment values) of ODI between control (16.60 ± 2.22) and study (26.50 ± 4.09) groups in two tailed unpaired t test, with α=0.05, power of 80%, and an effect size of 0.74. So, a sample size of 30 patients/per group would be required and increased to 35 women to allow for a 15% dropout rate (Power 301 http: www.psycho.uni-duesseldorf.de) Randomization. Randomization of sample selection were achieved using closed envelop way to allocate study participants to either intervention group (medication and treatment exercises) control group (medication only). all postmenopausal women and examiners were unaware of group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Their ages were ranged from 50-60 years.
* Their BMI not exceeded 30 kg/m2.
* All postmenopausal women past of at least one year after menopause.
* Had no regular physical activities during the past 6 months.

Exclusion Criteria:

* Patients didn't take any drug before the study (e.g. calcium tablets, multivitamins containing calcium and vitamin D) that affects bone metabolism.
* Patients that were smoking or having alcohol consumption.
* Histories of fracture and surgery, or severe injuries

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Dual-energy x-ray absorptiometry | period of treatment was 4 successive months.
  a valid and reliable method for assessing bone mineral density, A normal T score is -1.0 and above, low bone density is between -1.0 and -2.5, and osteoporosis is -2.5 and lower
Oswestry Disability Index | period of treatment was 4 successive months.
  reliable method for assessing quality of life, The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, standing, sleeping, sex life, social life and travelling.
  Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Emara, phd, Study Chair — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No